CLINICAL TRIAL: NCT05279573
Title: Randomized Controlled Intervention Study to Analyze the Efficacy of a Dietary Ingredient Combination With Omega-3 for Joint Function
Brief Title: Efficacy of a Dietary Ingredient Combination With Omega-3 for Joint Function
Acronym: 7DHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Collaborators: Evonik Operations GmbH (Unknown)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: UCAMCFE-00020
Record Dates: First submitted 2022-02-22; First posted 2022-03-15 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2021-11

CONDITIONS: Joint Function Disorder
Keywords: Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Combination of Omega-3 based product and botanical ingredient (Experimental): Consumption for 60 days. Subjects should consume two capsules in the morning and two capsules in the afternoon.
  Interventions: Dietary Supplement: Omega-3 and/or botanical ingredient
- Omega-3 based product (Experimental): Consumption for 60 days. Subjects should consume two capsules in the morning and two capsules in the afternoon.
  Interventions: Dietary Supplement: Omega-3 and/or botanical ingredient
- Botanical ingredient (Experimental): Consumption for 60 days. Subjects should consume two capsules in the morning and two capsules in the afternoon.
  Interventions: Dietary Supplement: Omega-3 and/or botanical ingredient
- Control group (Placebo Comparator): Consumption for 60 days. Subjects should consume two capsules in the morning and two capsules in the afternoon.
  Interventions: Other: Control product consumption

INTERVENTIONS:
Dietary Supplement: Omega-3 and/or botanical ingredient — Consumption for 60 days. Subjects should consume two capsules in the morning and two capsules in the afternoon.
  Arms: Botanical ingredient; Combination of Omega-3 based product and botanical ingredient; Omega-3 based product
Other: Control product consumption — Product with identical characteristics to the experimental product. Consumption for 60 days. Subjects should consume two capsules in the morning and two capsules in the afternoon.
  Arms: Control group

SUMMARY:
Randomized, controlled, double-blind intervention study of four parallel branches depending on the product consumed, to analyze the efficacy of an Omega-3 based product on the mobility and functionality of the evaluated joint.

DETAILED DESCRIPTION:
The duration of the study will be 60 days (8 weeks). Each day they will have to consume the product under investigation. Subjects who meet the selection criteria will be randomized into each of the study groups (A, B, C o D, depending on the group in which they have been randomized). Each day the subjects will have to fill in a diary regarding pain and concomitant medication.

They will make a total of two visits to the research laboratory and will perform the tests pre-established in the protocol. In addition, a follow-up telephone call will be made after 30 days of consume. Subsequently, a statistical analysis will be performed with the variables measured in the study to obtain the results.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (age: 40-75 YO).
* Subjects must have persistent knee pain with a baseline VAS pain assessment score of at least 30 mm.
* Subjects should not present narcotic drugs or steroidal anti-inflammatory drugs or immunosuppressants in their treatment.

Exclusion Criteria:

* Serious or terminal illnesses.
* Subjects currently taking glucosamine, chondroitin sulfate, collagen or hyaluronic infiltrations or any supplement indicated for joint health.
* Subjects who are currently consuming or have consumed in the last two months any Omega-3 based supplement and/or supplement based on the botanical ingredient under investigation.
* Subjects with chronic inflammatory diseases that affect the musculoskeletal system (rheumatoid arthritis, gout, pseudo-gout, Paget's disease, chronic pain syndrome, etc.).
* Subjects with a body mass index above 32.
* Subjects with known allergy to any of the study components.
* Pregnant or lactating women.
* Inability to understand informed consent.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Change in Pain from baseline at 8 weeks | The evolution of pain after consumption during 8 weeks will be measured.
  Visual analog scale from 0 to 10. The higher the value, the more pain.
Quality of life test: WOMAC test | Change in initial quality of life at 8 weeks.
  The quality of life of the subjects will be measured with the WOMAC test. It is a 24-item test that will measure the degree of pain: nothing, little, enough and a lot, when performing activities in daily life.

SECONDARY OUTCOMES:
Change in Pain from baseline at 8 weeks | Pain will be measured with a daily scale, from baseline to 8 weeks.
  Visual analog scale from 0 to 10. The higher the value, the more pain.
Functional test | The test will be measured at baseline and after 8 weeks of consumption.
  The balance and mobility of the subjects will be measured with the Timed Up and Go Test
Muscle function | The test will be measured at baseline and after 8 weeks of consumption.
  Isokinetic and isometric dynamometry
Change in concomitant analgesic medication | The test will be measured at baseline and after 8 weeks of consumption. It will also be evaluated on a daily basis
  The change in the need for the use of analgesic medications will be evaluated
Sleep efficiency | The test will be measured at baseline and after 8 weeks of consumption. It will be measured during 3 weekdays and one weekend day.
  Measured by accelerometry, with Actigraph wGT3X-BT
Sleep quality | It will be measured twice, once at baseline or at the end of the study after 8 weeks of use
  Measured by Pittsburgh test
Omega-3 Bioavailability | It will be measured twice, once at baseline or at the end of the study after 8 weeks.
  Measured by omega quant
Liver safety variables | It will be measured twice, once at baseline or at the end of the study after 8 weeks.
  It is a blood test that measures the presence of some enzymes, proteins and bilirubin in the blood, with the aim of determining if there is any alteration in the liver. Enzyme GPT, GOT, Gamma GT, LDH, alkaline phosphatase and bilirubin (UI/L)
Physical activity | The test will be measured at baseline and after 8 weeks of consumption. It will be measured during 3 weekdays and one weekend day.
  It is a control variable. Measured by accelerometry, with Actigraph wGT3X-BT
Physical activity control | The test will be measured at baseline and after 8 weeks of consumption.
  It is a control variable. Measured by fitbit
Body composition | The test will be measured at baseline and after 8 weeks of consumption.
  It is a control variable. Measured by bioimpedance
Waist - hip circumference | The test will be measured at baseline and after 8 weeks of consumption.
  It is a control variable.

CONTACTS AND LOCATIONS:
Overall Officials: Fco Javier López Roman, Principal Investigator — Catholic University of Murcia
Locations (1):
- Catholic University of Murcia, Murcia, Spain